CLINICAL TRIAL: NCT04829552
Title: Prophylactic Versus Therapeutic Dose Anticoagulation In COVID-19 Infection at the Time of Admission To Critical Care Units: A Multicenter Retrospective Cohort Study in the Beaumont Healthcare System
Brief Title: Prophylactic Versus Therapeutic Dose Anticoagulation In COVID-19 Infection at the Time of Admission To Critical Care Units
Status: Completed | Type: Observational
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Faisal Musa, MD, Staff Physician, Corewell Health East
Other Study IDs: 2020-219
Record Dates: First submitted 2021-03-22; First posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Covid19
Keywords: anticoagulation; COVID19; thrombosis; heparin; coagulopathy
MeSH Terms: conditions — COVID-19; Thrombosis; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: low dose group.: patients treated with subcutaneous low molecular weight heparin 40 mg once daily or unfractionated heparin 5000 IU twice or three times daily for at least 5 days.
- Study group: high dose group.: Patients treated with subcutaneous low molecular weight heparin 1 mg/kg twice daily or 1.5 mg/kg daily or a continuous intravenous infusion of unfractionated heparin for at least 5 days.

SUMMARY:
This is a multi-center, retrospective, study to determine if therapeutic dose anticoagulation (High dose group) improves inpatient mortality in severely ill patients with COVID-19 compared to prophylactic dose anticoagulation (Low dose group). The study involved 704 individuals who were admitted to Beaumont Health System (BHS) from March 10th to April 15th, 2020.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* positive reverse transcription-polymerase chain reaction (rRT-PCR) test for the qualitative detection of nucleic acid from SARS-CoV-2 in upper and lower respiratory specimens.
* Intensive care unit (ICU) patient or Step-down unit (SDU) patient on invasive mechanical ventilation, BiPAP, 100% non-rebreather mask, or high flow oxygen or supplemental oxygen of at least 4 liters per minute nasal cannula.
* peak d-dimer levels exceeding 1,000 mcg/mL at any time during admission.

Exclusion Criteria:

* Hospital length of stay less than 5 days.
* Hemorrhage before ICU/SDU admission.
* Treatment with an anticoagulant other than low molecular weight heparin or unfractionated heparin.
* Constant treatment with the same dose of anticoagulant for less than 5 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who were admitted to Beaumont Health System (Michigan, USA) ICU/SDU in the period of March 10th to April 15th, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 704 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Inpatient all-cause mortality | During hospitalization, up to 6 months

SECONDARY OUTCOMES:
Rates of major bleeding events | During hospitalization, up to 6 months
  as defined by the International Society on Thrombosis and Hemostasis
Rates of venous thromboses | During hospitalization, up to 6 months
Intensive care unit/Step down unit length of stay | During hospitalization, up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beaumont Health System (BHS), Royal Oak, Michigan, United States